CLINICAL TRIAL: NCT03510897
Title: A Randomized, Double-Blind, Placebo Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of QPI-1002 for the Prevention of Major Adverse Kidney Events (MAKE) in Subjects at High Risk for Acute Kidney Injury (AKI) Following Cardiac Surgery
Brief Title: QPI-1002 Phase 3 for Prevention of Major Adverse Kidney Events (MAKE) in Subjects at High Risk for AKI Following Cardiac Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study completed day 90 for primary endpoint but was terminated early for one year follow up due to results not meeting efficacy outcome at Day 90.
Sponsor: Quark Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: QRK309
Record Dates: First submitted 2018-04-18; First posted 2018-04-27 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Cardiac Surgery
Keywords: MAKE; AKI

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- QPI-1002 (Active Comparator): QPI-1002 Injection, Single dose
  Interventions: Drug: teprasiran
- Placebo (Placebo Comparator): isotonic saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: teprasiran — IV injection
  Other Names: QPI-1002
  Arms: QPI-1002
Drug: Placebo — isotonic saline
  Arms: Placebo

SUMMARY:
This trial is designed to evaluate QPI-1002 versus placebo for the prevention of Major Adverse Kidney Events (MAKE) in subjects at high risk for acute kidney injury following cardiac surgery. Half of the participants will receive QPI-1002 while the other half will receive placebo.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, Phase 3 trial to evaluate QPI-1002 versus placebo for the prevention of Major Adverse Kidney Events in subjects at high risk for acute kidney injury following cardiac surgery. Subjects will be dosed with active drug or placebo after the completion of cardiovascular surgery.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female, age ≥ 18 years old
* At risk for AKI following cardiac surgery on the basis of at least one of the following pre-operatively assessed risk factors:

  * Reduced renal function
  * Diabetes with ongoing insulin treatment
  * Albuminuria
* Undergoes non-emergent open chest cavity cardiovascular surgeries, with use of cardiopulmonary bypass (CPB), with or without hypothermic circulatory arrest

Key Exclusion Criteria:

* Emergent surgeries, including aortic dissection, and major congenital heart defects
* Undergoes cardiac surgery off CPB for subjects ≥45 years old. (Cardiac surgery off CPB for subjects <45 years old is allowed.)
* Perioperative or post cardiac surgery, an left ventricular assist device (LVAD) is inserted or anticipated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1043 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects through day 90 who develop major adverse kidney events | Baseline through day 90

SECONDARY OUTCOMES:
Proportion of subjects developing AKI overall by modified AKIN criteria within 5 days post-surgery | Baseline through day 5
Renal function as estimated by glomerular filtration rate | Baseline through Day 90
Proportion of subjects who die or initiate dialysis through day 90 | Baseline through day 90

CONTACTS AND LOCATIONS:
Overall Officials: Nitsan Halevy, MD, Study Director — Quark Pharmaceuticals
Locations (104):
- United States (36):
  - University of Alabama at Birmingham Hospital, Birmingham, Alabama
  - Keck Hospital of USC, Los Angeles, California
  - Cedar-Sinai Heart Institute, Los Angeles, California
  - Ronald Regan UCLA Medical Center, Los Angeles, California
  - Yale University School of Medicine, New Haven, Connecticut
  - River City Clinical Research, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northwestern University, Evanston, Illinois
  - Indiana/ Ohio Heart, a division of Luthern Medical Group, LLC, Fort Wayne, Indiana
  - Indiana University Health-Methodist Hospital, Indianapolis, Indiana
  - University of Kentucky Healthcare, Lexington, Kentucky
  - University of Louisville Physicians (ULP), Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - MidMichigan Medical Center Midland, Midland, Michigan
  - Cardiac & Vascular Research Center of Northern Michigan, Petoskey, Michigan
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Bryan Heart, Lincoln, Nebraska
  - Nebraska Heart Hospital, Lincoln, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Columbia University Medical Center, New York, New York
  - Mission Hospital, Inc., Asheville, North Carolina
  - Duke University Hospital Medical Center, Durham, North Carolina
  - East Carolina Heart Institute at East Carolina University, Greenville, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor Jack and Jane Hamilton Heart and Vascular Hospital - Soltero Cardiovasular, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah Health, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - University Hospital, Madison, Wisconsin
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Australia (9):
  - Westmead Hospital, Westmead, New South Wales
  - The Prince Charles Hospital, Chermside, Qeensland
  - Princess Alexandra Hospital, Woolloongabba, Qeensland
  - The Townsville Hospital, Douglas, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - St. Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Austria (3):
  - Medizinische Universitat Innsbruck, Innsbruck, Tyrol
  - Kepler Universitatsklinikum GmbH, Linz, Upper Austria
  - Medizinische Universitat Wien, Vienna
- University Hospital Leuven, Campus Gasthuisberg, Leuven, Belgium
- Canada (12):
  - Foothills Medical Centre, Libin Cardiovascular Institute of Alberta, University of Calgary, Calgary, Alberta
  - University of Alberta Hospital / Mazankowski Alberta Heart Institute, Edmonton, Alberta
  - Royal Jubilee Hospital (Victoria Island Health Authority), Victoria, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Horizon Health Network, Saint John Regional Hospital, Saint John, New Brunswick
  - Hamilton General Hospital, Hamilton, Ontario
  - London Health Sciences Center, University Hospital, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - McGill University Health Center - Royal Victoria Hospital, Montreal, Quebec
  - Institut Universitaire de cardiologie et de pneomologie de Quebec, Universite Laval, Québec, Quebec
- Czechia (3):
  - Fakulni nemocnice Hradec Kralove, Kardiochirurgicka klinika, Hradec Králové
  - Institut klinicke a experimenalni mediciny, Klinika kardiovaskularni chirurgie, Prague
  - Fakultni nemocnice Motol a 2. LF UK, Klinika kariovaskularni chirurgie 2. LF. UK, Prague
- France (7):
  - CHU Besancon-Service de Chirurgie Thoracique et Cardiovasculaire, Besançon
  - CHU - Grenoble Alpes, Grenoble
  - CHU Bordeaux, Pessac
  - Hospital Robert Debre, Reims
  - Chu Pontchaillou Rennes, Rennes
  - Hopitaux Universitaires de Strasbourg - Service de Chirurgie Cardiovasculaire, Strasbourg
  - CHU Toulouse - Hospital Rangueil-Service de Chirurgie Cadriovasculaire, Toulouse
- Germany (18):
  - Deutsches Herzzentrum Munchen, München, Bavaria
  - Charite-Universitatsmedizin Berlin, Berlin, Brandenburg
  - Klinikum der Friedrich-Schiller-Universitat Jena, Jena, Deutschland
  - Universitatsklinikum Frankfurt am Main, Frankfurt am Main, Hesse
  - Universitasklinikum Giessen und Marburg GmbH, Geißen, Hesse
  - Herz-Und Gefasszentrum Bad Bevensen, Bad Bevensen, Lower Saxony
  - Krankenhaus der Barmherzigen Bruder Trier, Trier, Rhineland-Palatinate
  - Herzzentrum Leipzig, Leipzig, Saxony
  - Universitats-Herzzentrum Freiburg-Bad Krozingen, Bad Krozingen
  - RHON-KLINIKUM Campus Bad Neustadt, Bad Neustadt an der Saale
  - Deutsches Herzzentrum Berlin, Berlin
  - Universitatsklinikum Bonn, Bonn
  - Universitatsklinikum "Carl Gustav Carus" der Technischen Universitat Dresden Klinik fur Herzchirurgle, Dresden
  - Universitatklinicum Essen Westdeutsches Herzzentrum Essen, Essen
  - Universitatsklinikum Heidelberg und Medizinische Fakultat, Heidelberg
  - Universitatsklinikum Schleswig-Holstein, Campus Lubeck, Lübeck
  - Universitatsmedizin der Johannes Gutenberg-Universitat Mainz, Mainz
  - Herzchirurgische Klinik und Poliklinik, München
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Waikato Hospital, Hamilton
  - Wellington Regional Hospital, Wellington
- Spain (10):
  - Hospital Clinico Universitario de Santiago-CHUS, Santiago de Compostela, A Coruña
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba, Cordoba
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Universitario de Cruces, Barakaldo
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Clinic Universitario de Valencia, Valencia
- United Kingdom (2):
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge, Cambridgeshire
  - Guy's and St Thomas Hospital, London

REFERENCES:
- [Derived] Scurt FG, Bose K, Mertens PR, Chatzikyrkou C, Herzog C. Cardiac Surgery-Associated Acute Kidney Injury. Kidney360. 2024 Jun 1;5(6):909-926. doi: 10.34067/KID.0000000000000466. Epub 2024 May 1. PMID 38689404
- [Derived] Thielmann M, Corteville D, Szabo G, Swaminathan M, Lamy A, Lehner LJ, Brown CD, Noiseux N, Atta MG, Squiers EC, Erlich S, Rothenstein D, Molitoris B, Mazer CD. Teprasiran, a Small Interfering RNA, for the Prevention of Acute Kidney Injury in High-Risk Patients Undergoing Cardiac Surgery: A Randomized Clinical Study. Circulation. 2021 Oct 5;144(14):1133-1144. doi: 10.1161/CIRCULATIONAHA.120.053029. Epub 2021 Sep 3. PMID 34474590
- [Derived] Hinze C, Karaiskos N, Boltengagen A, Walentin K, Redo K, Himmerkus N, Bleich M, Potter SS, Potter AS, Eckardt KU, Kocks C, Rajewsky N, Schmidt-Ott KM. Kidney Single-cell Transcriptomes Predict Spatial Corticomedullary Gene Expression and Tissue Osmolality Gradients. J Am Soc Nephrol. 2021 Feb;32(2):291-306. doi: 10.1681/ASN.2020070930. Epub 2020 Nov 25. PMID 33239393